CLINICAL TRIAL: NCT00162084
Title: A Phase 3, Parallel, Double Blind, Multicenter Trial to Examine Inducible Myocardial Perfusion Abnormality Detection With BMS068645 and Adenosine Stress SPECT Compared to Coronary Angiography
Brief Title: A Study to Examine MPI SPECT Imaging With BMS068645 and Adenosine Compared to Coronary Angiography
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision to stop the program
Sponsor: Forest Laboratories (Industry)
Responsible Party: Amy Lankford, PhD, Sr. Manager, PGxHealth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: BMS068645-302
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Heart Disease; Ischemic Heart Disease
MeSH Terms: conditions — Heart Diseases; Myocardial Ischemia

INTERVENTIONS:
Drug: apadenoson

SUMMARY:
The purpose of the study is to determine whether BMS068645 is as effective as Adenosine SPECT at detecting blockages in heart arteries, and to determine if it will have fewer side effects

ELIGIBILITY:
Inclusion Criteria:

* Referral for pharmacologic stress SPECT MPI
* Have suspected Ischemic heart disease

Exclusion Criteria:

* Acute myocardial Infarction, Coronary artery bypass graft, percutaneous coronary intervention within 30 days of enrollment
* Severe asthma or COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 2005-04; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of BMS068645 vs. adenosine; to be determined at the end of the study after enrollment is complete

SECONDARY OUTCOMES:
Incidence of serious adverse events due to adenosine vs. BMS068645; incidence of adverse events due to adenosine vs. BMS068645; to be determined at the end of the study after enrollment, but with interim independent analysis by a safety monitoring board

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hibberd, MD, PhD, Study Director — Bristol-Myers Squibb
Locations (72):
- United States (72):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Huntsville, Alabama
  - Local Institution, North Little Rock, Arkansas
  - Local Institution, Northridge, California
  - Local Institution, Rancho Mirage, California
  - Local Institution, Santa Clara, California
  - Local Institution, Santa Rosa, California
  - Local Institution, Walnut Creek, California
  - Local Institution, Bridgeport, Connecticut
  - Local Institution, Guilford, Connecticut
  - Local Institution, New Haven, Connecticut
  - Local Institution, Newark, Delaware
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Gainesville, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Jacksonville Beach, Florida
  - Local Institution, Jupiter, Florida
  - Local Institution, Miami, Florida
  - Local Institution, Safety Harbor, Florida
  - Local Institution, Stuart, Florida
  - Local Institution, Tamarac, Florida
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Aurora, Illinois
  - Local Institution, Fox River Grove, Illinois
  - Local Institution, La Grange, Illinois
  - Local Institution, Peoria, Illinois
  - Local Institution, Winfield, Illinois
  - Local Institution, Fort Wayne, Indiana
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Overland Park, Kansas
  - Local Institution, Louisville, Kentucky
  - Local Institution, Baton Rouge, Louisiana
  - Local Institution, Auburn, Maine
  - Local Institution, Scarborough, Maine
  - Local Institution, South Portland, Maine
  - Local Institution, Westminster, Maryland
  - Local Institution, Ayer, Massachusetts
  - Local Institution, Grand Rapids, Michigan
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, Saint Cloud, Minnesota
  - Local Institution, Saint Louis Park, Minnesota
  - Local Institution, Tupelo, Mississippi
  - Local Institution, Kansas City, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Albany, New York
  - Local Institution, New York, New York
  - Local Institution, West Islip, New York
  - Local Institution, Raleigh, North Carolina
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Cleveland, Ohio
  - Local Institution, Columbus, Ohio
  - Local Institution, Lorain, Ohio
  - Local Institution, Sandusky, Ohio
  - Local Institution, Westlake, Ohio
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Wyomissing, Pennsylvania
  - Local Institution, Providence, Rhode Island
  - Local Institution, Simpsonville, South Carolina
  - Local Institution, Chattanooga, Tennessee
  - Local Institution, Johnson City, Tennessee
  - Local Institution, Nashville, Tennessee
  - Local Institution, Oak Ridge, Tennessee
  - Local Institution, Amarillo, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Plano, Texas
  - Local Institution, Hopewell, Virginia
  - Local Institution, Lynchburg, Virginia
  - Local Institution, Richmond, Virginia
  - Local Institution, Roanoke, Virginia
  - Local Institution, Spokane, Washington
  - Local Institution, Wausau, Wisconsin